CLINICAL TRIAL: NCT04869163
Title: Sustained Wellbeing Benefits of Red Meat Consumption in a Modern Flexitarian Diet: A Study Protocol for a 10 Week Randomised Clinical Trial
Brief Title: Sustained Meat and Alternative Intake (PRotEin DIet SatisfacTION Trial 4) (PREDITION)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: AgResearch (Unknown); University of Otago (Other)
Responsible Party: Principal Investigator, Dr Andrea Braakhuis, Principal Investigator, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5000927-4
Record Dates: First submitted 2021-04-18; First posted 2021-05-03 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Well-being
Keywords: nutrition; meat; mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- red meat consumers (Active Comparator): Consumes red meat 3 times a week
  Interventions: Other: Non-red meat
- non-red meat consumers (Experimental): Consumes a non-red meat comparison product 3 times a week
  Interventions: Other: Non-red meat

INTERVENTIONS:
Other: Non-red meat — Red meat analogues and alternatives

SUMMARY:
Introduction The trend of flexitarian eating patterns is on the rise, with young adults amongst the biggest adopters claiming health and environmental reasons to reduce red meat intake. Nutrient dense meat and animal products are often the lynchpin of these diets, even when consumed only occasionally and in moderate amounts. Red meat provides forms and concentrations of essential proteins, lipids, and micronutrients that are scarce in exclusively vegetarian regimens. The aim of this investigation is to consider the effects of moderate consumption of lean red meat as part of an otherwise vegetarian balanced diet and its impact on biomarkers of sustained health and wellbeing.

Methods and analyses A cohort of healthy, young (20-34 years) male and female participants will take part in two-arm parallel, randomised-controlled trial for a duration of 12 weeks, with a 3-month post follow-up. The trial will commence with a two-week assessment period followed by allocation to the intervention arms. The intervention will include the consumption of red meat or meat-alternatives three times per week for 10 weeks. Blood samples of the participants will be measured for changes in erythrocyte fatty acid distribution, circulating amino acids, neurotransmitters, markers of mineral status and inflammatory markers. Questionnaires to assess wellbeing and mental health will be undertaken every two weeks. Body composition, physical function test, blood measurements will be assessed at allocation (t0), week five into the intervention (t5) and post intervention (t10).

Discussion To our knowledge this is the first randomised controlled trial (RCT) investigating the overarching health consequences of consuming NZ pasture fed red meat or no meat, as part of a healthy diet.

Ethics and dissemination The trial was approved by the New Zealand Ministry of Health's Health and Disability Ethics Committees (20/STH/157).

DETAILED DESCRIPTION:
Study Design and Setting The study is a parallel RCT comprising a 2-week pre-intervention assessment, a 10-week intervention period and a 22-week post follow up. Participants will all eat a balanced plant-based basal diet and be randomised to also consume either red meat ('Flexitarian' arm) or a meat substitute ('Vegetarian' arm). The meat will be pasture-raised beef and lamb butchered and packaged to our specifications in New Zealand, while the meat substitute will be commercially available plant-based products.

Recognising that there are many interpretations of the terms vegetarian and flexitarian, in this study we define vegetarian as ovo-lacto vegetarian and flexitarian as 'a vegetarian diet with moderate amounts of red meat'. Both arms can consume eggs and dairy products, but no chicken, pork or fish, and no red meat other than that supplied by the researchers.

The study is designed around pairs of young adult consumers who share meals and are therefore likely to engage over the values and challenges of developing a healthy lifestyle. Each couple/household unit (see Recruitment) will receive a weekly delivery of a vegetarian meal kit containing complete ingredients for cooking 3-4 evening meals. Depending on their allocation, the couple will also receive an allotment of frozen red meat or meat-analogue to use for preparing 3 additional evening meals. To facilitate cooking and keep the behaviours of the arms aligned, we will provide recipe cards, shopping guidance and video instructions. All other meals during the week are self-catered and must adhere to study guidelines.

The quantity of meat will be sufficient to provide 350-500 g cooked weight per person per week. This conforms to the latest international recommendations for maximum intake 7 and the reported typical frequencies of red meat consumption. The meat alternative will be similar in quantity, form and function. It is vegetarian-friendly and serves to balance the total protein and fat intake of the arms.

Changes in objective and self-assessed subjective health variables over time and between arms will be investigated. These include physical function, body composition, metabolic health biomarkers and psychological wellbeing.

ELIGIBILITY:
Inclusion criteria:

* All participants are required to be omnivores who in the last 2 months consumed at least 2-3 meals per week containing meat of any description (red or white fleshed meat, including fish).
* All participants must be willing to consume both red meat and meat-analogues for the purposes of the trial.

Exclusion criteria:

* Obesity (BMI ≥ 30 kg/m2),
* Hyperlipidaemia
* Anosmia and ageusia (issues with smell and taste),
* Use of medications (except for occasional NSAIDs and antihistamines) or recreational drugs, or who smoke tobacco
* Disordered eating

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Polyunsaturated fatty acids | Baseline to 10 week comparison
  Concentrations of polyunsaturated fatty acids (18:2 n-6, 18:3 n-3, 20:4 n-6, 20:5 n-3, 22:5 n-3, 22:6 n-3) in erythrocyte membranes

SECONDARY OUTCOMES:
Psychological and mental wellbeing | Change from baseline to 10 week comparison
  Multidimensional Fatigue Symptom Inventory Short Form (MSFI-SF). The Total MFSI-SF score ranges from -24 to 96, with higher values indicating greater fatigue.
  The five subscales of the MFSI each ranges from 0 to 24:
  1. General subscale = ranges from 0 to 24, with higher values indicating greater fatigue (worse outcomes)
  2. Physical subscale = ranges from 0 to 24, with higher values indicating greater fatigue (worse outcomes)
  3. Emotional subscale = ranges from 0 to 24, with higher values indicating greater fatigue (worse outcomes)
  4. Mental subscale = ranges from 0 to 24, with higher values indicating greater fatigue (worse outcomes)
  5. Vigor subscale = ranges from 0 to 24, with higher values indicating greater vigor (better outcomes) Total MFSI-SF score = (General + Physical + Emotional + Mental) - Vigor = Total Score ranges from -24 to 96 with higher values indicating greater fatigue (worse outcomes).
Psychological and mental wellbeing | Change from baseline to 10 week comparison
  Depression Anxiety Stress Scales-Short form (DASS-21) Depression score ranges from 0 to 42 (raw scores 0 to 21, which are then multiplied by 2 to be equivalent to the DASS-42), with higher numbers indicating greater depression (worse outcome).
  Anxiety score ranges from 0 to 42 (raw scores 0 to 21, which are then multiplied by 2 to be equivalent to the DASS-42), with higher numbers indicating greater anxiety (worse outcome).
  Stress score ranges from 0 to 42 (raw scores 0 to 21, which are then multiplied by 2 to be equivalent to the DASS-42), with higher numbers indicating greater stress (worse outcome).
Psychological and mental wellbeing | Change from baseline to 10 week comparison
  WHO-Five Well-Being Index (WHO 5). The raw score ranges from 0 to 25, with 0 representing the worst and 100 representing the best possible quality of life The percentage score ranges from 0 to 100, with 0 representing the worst and 100 representing the best possible quality of life
Psychological and mental wellbeing | Change from baseline to 10 week comparison
  Positive Eating Scale (PES) Total Positive Eating score (PES-Tot) = ranges from 1 to 4, with higher values indicating better experiences with eating Satisfaction with Eating subscale (PES-Sat) = ranges from 1 to 4, with higher values indicating more satisfaction with eating Pleasure when Eating subscale (PES-Pl) = ranges from 1 to 4, with higher values indicating more pleasure when eating

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Auckland, Auckland, [other], New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Access to data will be granted to appropriate members of the research team and to authorised representatives from the host institution to monitor or audit the study and ensure compliance with regulations. Data will be made available to external academics on reasonable request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be made available when he study is complete (July 2022)

REFERENCES:
- [Derived] Worthington A, Gillies N, Hannaford R, Roy R, Braakhuis A. Implementing multicomponent, eHealth-based behaviour change support within a dietary intervention trial improves adherence to study-related behaviours in healthy young adults. BMC Nutr. 2023 Nov 21;9(1):134. doi: 10.1186/s40795-023-00798-7. PMID 37990250
- [Derived] Gillies NA, Worthington A, Li L, Conner TS, Bermingham EN, Knowles SO, Cameron-Smith D, Hannaford R, Braakhuis A. Adherence and eating experiences differ between participants following a flexitarian diet including red meat or a vegetarian diet including plant-based meat alternatives: findings from a 10-week randomised dietary intervention trial. Front Nutr. 2023 Jun 14;10:1174726. doi: 10.3389/fnut.2023.1174726. eCollection 2023. PMID 37388633
- [Derived] Braakhuis A, Gillies N, Worthington A, Knowles S, Conner T, Roy R, Pham T, Bermingham E, Cameron-Smith D. A Modern Flexitarian Dietary Intervention Incorporating Web-Based Nutrition Education in Healthy Young Adults: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Dec 21;10(12):e30909. doi: 10.2196/30909. PMID 34931994

DOCUMENTS (1):
  • Informed Consent Form (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT04869163/ICF_000.pdf